CLINICAL TRIAL: NCT01767324
Title: Exploratory Evaluation of Injection Sites in Healthy Subjects Receiving Saline Delivered by a Non-Significant Risk Investigational Device Utilizing a Micro-Needle Array
Brief Title: Site Selection for Intracutaneous Saline Delivery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: FluGen Inc (Industry)
Collaborators: Accelovance (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: FGN-NSR-2012-001
Record Dates: First submitted 2013-01-09; First posted 2013-01-14 (Estimated); Last update posted 2017-08-02 (Actual); Status verified 2017-07

CONDITIONS: Intracutaneous Drug Delivery
Keywords: microneedle-based array; hollow microneedle; intracutaneous; drug delivery; vaccine delivery

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Injection to deltoid (Experimental): Deliver saline from FLUGEN 101.2 microneedle-based delivery device.
  Interventions: Device: Injection to deltoid
- Injection to forearm (Experimental): Deliver saline from FLUGEN 101.2 microneedle-based delivery device.
  Interventions: Device: Injection to forearm
- Injection to thigh (Experimental): Deliver saline from FLUGEN 101.2 microneedle-based delivery device.
  Interventions: Device: Injection to thigh

INTERVENTIONS:
Device: Injection to deltoid — Deliver 0.5 milliliters of saline intradermally
  Arms: Injection to deltoid
Device: Injection to forearm — Deliver 0.5 milliliters of saline intradermally
  Arms: Injection to forearm
Device: Injection to thigh — Deliver 0.5 milliliters of saline intradermally
  Arms: Injection to thigh

SUMMARY:
The goal of this exploratory study is to select the optimal body site for intracutaneous delivery of 0.5 milliliters of saline from the FLUGEN 101.2 microneedle-based device.

DETAILED DESCRIPTION:
Test ability to inject saline into various sites on body.

ELIGIBILITY:
Inclusion Criteria:

* Able to read and/or understand and sign the Informed Consent Form

Exclusion Criteria:

* Medical history of acute or chronic skin disease
* Active skin allergy or acute skin infection, tattoo(s), scars, sunburn or skin abnormalities at any prospective injection site
* Hirsute at any prospective injection site
* Diabetes
* High levels of anxiety or depression or history of psychosis
* Abuse of alcohol or use of other drugs of abuse including tobacco
* Pregnant or breastfeeding women
* Any medical condition that may interfere with study protocol adherence including completion of study activities
* Foreseeable inability to complete the study as scheduled.

Ages: 18 Years to 49 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2012-12; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
The primary objective is to evaluate the safety and tolerability/reactogenicity of saline delivery from the FLUGEN 101.2 microneedle-based device as evidenced by change of dose site appearance over time. | 30 minutes, 24 hours, 1 week
  Observe injection sites for change of appearance post-dose including wheal formation or resolution.

SECONDARY OUTCOMES:
A secondary objective of this study is to evaluate the mechanical elimination of fluid from the device. | 3 minutes
  Evaluate ability of device to dispense targeted dose volume.

CONTACTS AND LOCATIONS:
Overall Officials: Renee Herber, Study Director — FluGen Inc; Murray A Kimmel, DO, Principal Investigator — Accelovance
Locations (1):
- Accelovance Inc, Melbourne, Florida, United States